CLINICAL TRIAL: NCT07231211
Title: An Open-label, Multicenter Phase I/II Clinical Study of SHR-4610 Injection in Patients With Advanced Solid Tumors to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy
Brief Title: A Study of SHR-4610 Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4610-101
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 Group (Experimental): SHR-4610 dose A in dose escalation stage.
  Interventions: Drug: SHR-4610 Injection
- Cohort 2 Group (Experimental): SHR-4610 dose B in dose escalation stage.
  Interventions: Drug: SHR-4610 Injection
- Cohort 3 Group (Experimental): SHR-4610 dose C in dose escalation stage.
  Interventions: Drug: SHR-4610 Injection
- Cohort 4 Group (Experimental): SHR-4610 dose D in dose escalation stage.
  Interventions: Drug: SHR-4610 Injection
- Cohort 5 Group (Experimental): SHR-4610 dose A/B/C/D in dose expansion stage.
  Interventions: Drug: SHR-4610 Injection
- Cohort 6 Group (Experimental): SHR-4610 dose A/B/C/D in efficacy expansion stage.
  Interventions: Drug: SHR-4610 Injection

INTERVENTIONS:
Drug: SHR-4610 Injection — SHR-4610 injection in different dose.

SUMMARY:
This study is an open, multicenter Phase I/II clinical trial, divided into two stages: dose exploration (including dose escalation and dose extension) and efficacy extension.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form;
2. Age range: 18-75 years old, both male and female are welcome;
3. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors which is relapsed or refractory to standard treatment, or lack of standard treatment;
4. Have at least one measurable tumor lesion per RECIST v1.1;
5. ECOG performance status of 0-1;
6. Life expectancy ≥ 12 weeks;
7. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Patients with active central nervous system metastases or meningeal metastases;
2. Systemic antitumor therapy was received 4 weeks before the start of the study;
3. Moderate or severe ascites with clinical symptoms; Uncontrolled or moderate or higher pleural effusion or pericardial effusion;
4. Have poorly controlled or severe cardiovascular disease;
5. Subjects with active hepatitis B or active hepatitis C;
6. Adverse reactions of previous anti-tumor treatment have not recovered to Grade ≤ 1 per NCI-CTCAE v5.0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Dose-Limiting Toxicity (DLT) | Post-dose at day 1 to the end of treatment visit, about 1 year.
The Maximum Tolerated Dose (MTD) | Post-dose at day 1 to the end of treatment visit, about 1 year.
Recommended dosage for Phase II (RP2D) | Post-dose at day 1 to the end of treatment visit, about 1 year.
Incidence and severity of adverse events (AEs) | Up to 90 days after the last administration.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the first administration to the end of treatment visit, about 1 year.
Duration of relief (DOR) | From the first administration to the end of treatment visit, about 1 year.
Disease Control Rate (DCR) | From the first administration to the end of treatment visit, about 1 year.
Time to Response (TTR) | From the first administration to the end of treatment visit, about 1 year.
Progression-free survival (PFS) | From the first administration to the end of treatment visit, about 1 year.
Time to the maximum plasma concentration (Tmax) | From Day 1 pre-dose to 30 days after the last administration.
Maximum concentration of SHR-4610 (Cmax) | From Day 1 pre-dose to 30 days after the last administration.
SHR-4610 serum trough concentration (Ctrough) | From Day 1 pre-dose to 30 days after the last administration.
Area under the concentration versus time curve of SHR-4610 from time zero to time t (AUC0-t) | From Day 1 pre-dose to 30 days after the last administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided